CLINICAL TRIAL: NCT01641432
Title: Computerized Cognitive Treatment of Vigilance Deficits in Individuals With Acquired Brain Injury
Brief Title: Computerized Attention Training for Individuals With Acquired Brain Injury
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Posit Science Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: BPI-1002-2011
Record Dates: First submitted 2012-06-25; First posted 2012-07-16 (Estimated); Last update posted 2014-07-22 (Estimated); Status verified 2014-07

CONDITIONS: Acquired Brain Injury; Stroke; Hemispatial Neglect
MeSH Terms: conditions — Brain Injuries; Stroke; Perceptual Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider

ARMS (2):
- TAPAT (Experimental): Computerized Tonic and Phasic Attention training consisting of visual, auditory, and spatial stimuli that requires sustained attention (24 minutes). Training is followed by a computerized cognitive exercise (12 minutes).
  Interventions: Behavioral: Tonic and Phasic Attention Training
- Active Comparator (Active Comparator): Computerized conventional board-games that lack the therapeutic effect of the TAPAT exercises. Active control has stimulus parameters similar to the TAPAT exercises (eg. stimuli is presented on the computer, participant responses are collected, session time and improvement is measured).
  Interventions: Behavioral: Active Comparator

INTERVENTIONS:
Behavioral: Tonic and Phasic Attention Training — The Tonic and Phasic Alertness treatment task (TAPAT) consist of two consecutive rounds of a 12-minute continuous performance task in which continually varying, rich visual (e.g., scenes, objects, faces) or auditory stimuli (tones or complex sounds) are briefly displayed and participants are required to respond via a button press when they see a non-target item (90% of trials) or withhold button-press responding when the item is a pre-determined target item (10% of trials). Presentation of the target item is non-predictive and infrequent, disallowing the development of an executive strategy. Participants simply sustain attention to the task over a prolonged period of time (tonic attention), ignoring distractions, and inhibiting the pre-potent motor response when they see a target item (phasic attention).
  Following the 24 minutes of TAPAT treatment participants will undergo one additional computer-based cognitive exercise, Multiple Object Tracking (MOT), for an additional 12 minutes.
  Arms: TAPAT
Behavioral: Active Comparator — Computer games chosen from a list of progressive visual/audiovisual games from the top-100 game list: sporcle.com. Training duration will be similar to that of experimental training.
  Arms: Active Comparator

SUMMARY:
Problems with attention are a common and debilitating consequence of brain injury. Studies show that poor attention is the number one predictor of poor cognitive functioning one year post-injury. This is due to the fact that attention is a necessary component of more complex cognitive functions such as learning & memory, multi-tasking and problem solving. In many cases, individuals may exhibit problems with spatial attention known as 'hemi-spatial neglect syndrome' or simply 'neglect'. Many studies now show that the processing machinery of the brain is plastic and remodeled throughout life by learning and experience, enabling the strengthening of cognitive skills or abilities. The investigators own research has shown that brief, daily computerized cognitive training that is sufficiently challenging, goal-directed and adaptive enables intact brain structures to restore balance in attention and compensate for disruptions in cognitive functioning.

DETAILED DESCRIPTION:
Participants will first engage in an assessment process to determine current level of cognitive function. This process consists of paper-pencil surveys and computerized tests. Following the assessment process, participants will engage in Internet browser-delivered training sessions conducted on any internet-accessible computer. These trainings can be done up to 7 times a week (once a day) or at participant's convenience (the investigators recommend 4-5 times a week). Following the completion of training, participant's cognitive function will be re-assessed. Participation is voluntary and participants may withdraw from the study at any time.

ELIGIBILITY:
Inclusion:

1. Participants must 21 years or older and not pregnant as indicated by self-report
2. Participant must be fluent in English (indicated by self-report)
3. Participant must be able to engage with computerized cognitive tasks as indicated by investigator's opinion after 30 minutes of computer interaction
4. Participants should have no history of chronic psychiatric or neurological condition (preceding the current insult) as indicated by self-report
5. Normal vision (or corrected to normal vision) as indicated by self-report
6. Participants must be willing to commit to the time requirements of the study as evidenced by written, informed consent.
7. Evidence of hemispatial neglect and/ or vigilance decline on at least one standard measure (e.g., A-SCAN).

Exclusion:

1. Participants report or present a hand tremor that prevents the use of a computer mouse or keyboard, in the opinion of the evaluating Principal or Sub-Investigator.
2. Unable to perform neuropsychological evaluations in the opinion of the evaluating Principal or Sub-Investigator.
3. In the opinion of the consenting staff person, the participant cannot comprehend, follow instructions, or is incapable of providing written, informed consent.
4. In the opinion of the consenting staff person, participant is not capable of giving informed consent and does not have a Legal Authorized Representative.
5. History of recurrent psychiatric impairment as indicated by self-report.
6. History of drug or alcohol abuse as indicated by self-report.
7. History of significant medical diseases or multiple neurological events of the head as indicated by self-report.

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2011-07; Primary Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Attention and Memory | 6 months
  Percent change on standardized measures of attention and executive function (all participants) using the ASCAN, Attentional Blink, Attention Capture Task, Landmark task, Conjunction Search task, SART, Verbal Fluency, CVLT-II, D-KEFS Stroop, and LNS assessments.

CONTACTS AND LOCATIONS:
Locations (1):
- Brain Plasticity Institute, San Francisco, California, United States